CLINICAL TRIAL: NCT00411983
Title: A Long-term Follow-up Study for HIV-infected Individuals Who Have Participated in HIV-NAT Study Protocols
Brief Title: A Long-term Follow-up of the HIV-NAT Cohort
Status: Recruiting | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT 006
Record Dates: First submitted 2006-12-14; First posted 2006-12-15 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections
Keywords: chronic HIV infection; long term cohort of HIV infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMC collection once a year
Oversight: Data Monitoring Committee: Yes

SUMMARY:
With HIV/AIDS increasingly considered a chronic disease, 24-, or 48-week data from antiretroviral studies are no longer sufficient. Only with long-term follow-up and outcome data will shed some much-needed light on the answers of questions that have stumped us for several years. Data from a large observational cohort of patients treated with combination antiretroviral therapy will provide further insights into the long-term safety and durability of various antiretroviral therapeutic approached, the efficacy of HIV viral load and CD4 cell counts as predictors of disease progression and mortality, and the importance of adherence.

DETAILED DESCRIPTION:
Primary Objective:

To collect and evaluate long-term clinical outcomes of HIV infected participants previously enrolled in HIV-NAT trials.

Secondary Objective:

To Assess:

1. Long-term consequences of initiation of antiretroviral as predicted by baseline CD4 cell count and/or baseline plasma HIV RNA level
2. Incidence of lipodystrophy and other metabolic complications in three different groups of patients initially treated with NRTI-based regimens, NNRTI-based regimens, or PI-based regimens
3. Class-specific incidence of lipodystrophy and metabolic complications such as d4T versus AZT, nevirapine versus efavirenz and individual PIs (IDV, SQV, Kaletra, and atazanavir)
4. Resistance profiles in patients on different antiretroviral regimens
5. Long-term consequences of antiretroviral agents on cardiovascular, renal, hepatic, and endocrine function, skin, gastrointestinal system and urogentital tract
6. Incidence of opportunistic infections or malignancy including hepatocarcinoma in patients with HIV/HCV or HIV/HBV co-infection
7. Immune recovery syndrome
8. Adherence to different antiretroviral regimens
9. Quality of life

ELIGIBILITY:
Inclusion Criteria:

* HIV infected patients( children and adults) previously participated HIV-NAT studies
* HIV infected patients( children and adults) currently participate in HIV-NAT trials
* Able to provide written consent

Exclusion Criteria:

* Unable to provide written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All HIV infected adult patients from HIV-NAT.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2002-11 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
HIV infection | 30 years
  This cohort will collect various information such as but not limited to:
  comorbidity, mortality, cardiovascular, neurological clinical data, treatment history, serious adverse events, PBMCs, clinical outcomes, virological outcomes, resistance, failure, aging, other opportunistic infections, etc

CONTACTS AND LOCATIONS:
Overall Officials: Praphan Phanuphak, MD, PhD, Principal Investigator — HIV-NAT, Thai Red Cross AIDS Research Center
Locations (1):
- HIV-NAT, Thai Red Cross AIDS Research Center, Bangkok, Thailand

REFERENCES:
- [Result] Law WP, Duncombe CJ, Mahanontharit A, Boyd MA, Ruxrungtham K, Lange JM, Phanuphak P, Cooper DA, Dore GJ. Impact of viral hepatitis co-infection on response to antiretroviral therapy and HIV disease progression in the HIV-NAT cohort. AIDS. 2004 May 21;18(8):1169-77. doi: 10.1097/00002030-200405210-00010. PMID 15166532
- [Result] Law WP, Dore GJ, Duncombe CJ, Mahanontharit A, Boyd MA, Ruxrungtham K, Lange JM, Phanuphak P, Cooper DA. Risk of severe hepatotoxicity associated with antiretroviral therapy in the HIV-NAT Cohort, Thailand, 1996-2001. AIDS. 2003 Oct 17;17(15):2191-9. doi: 10.1097/00002030-200310170-00007. PMID 14523276
- [Result] Avihingsanon A, Kerr SJ, Punyawudho B, van der Lugt J, Gorowara M, Ananworanich J, Lange JM, Cooper DA, Phanuphak P, Burger DM, Ruxrungtham K. Short communication: Aging not gender is associated with high atazanavir plasma concentrations in Asian HIV-infected patients. AIDS Res Hum Retroviruses. 2013 Dec;29(12):1541-6. doi: 10.1089/aid.2013.0069. Epub 2013 Oct 2. PMID 24088045
- [Result] Clarke A, Kerr S, Honeybrook A, Cooper DA, Avihingsanon A, Duncombe C, Phanuphak P, Ruxrungtham K, Ananworanich J, Kaldor J. Adherence and Risk Behaviour in Patients with HIV Infection Receiving Antiretroviral Therapy in Bangkok. Open Virol J. 2012;6:23-8. doi: 10.2174/1874357901206010023. Epub 2012 Feb 24. PMID 22423306
- [Result] Nuesch R, Srasuebkul P, Ananworanich J, Ruxrungtham K, Phanuphak P, Duncombe C; HIV-NAT Study Team. Monitoring the toxicity of antiretroviral therapy in resource limited settings: a prospective clinical trial cohort in Thailand. J Antimicrob Chemother. 2006 Sep;58(3):637-44. doi: 10.1093/jac/dkl313. PMID 16895939
- [Result] Avihingsanon A, Tongkobpetch S, Kerr SJ, Punyawudho B, Suphapeetiporn K, Gorowara M, Ruxrungtham K, Shotelersuk V. Pharmacogenetic testing can identify patients taking atazanavir at risk for hyperbilirubinemia. J Acquir Immune Defic Syndr. 2015 May 1;69(1):e36-7. doi: 10.1097/QAI.0000000000000540. No abstract available. PMID 25622064
- [Result] Kerr SJ, Punyawudho B, Thammajaruk N, Colbers A, Chaiyahong P, Phonphithak S, Sapsirisavat V, Ruxrungtham K, Burger DM, Avihingsanon A. Factors associated with daily tenofovir exposure in Thai subjects taking combination antiretroviral therapy. AIDS Res Hum Retroviruses. 2015 Apr;31(4):368-74. doi: 10.1089/AID.2014.0249. Epub 2014 Dec 17. PMID 25384393
- [Result] Avihingsanon A, Ramautarsing RA, Suwanpimolkul G, Chetchotisakd P, Bowonwatanuwong C, Jirajariyavej S, Kantipong P, Tantipong H, Ohata JP, Suankratay C, Ruxrungtham K, Burger DM. Ergotism in Thailand caused by increased access to antiretroviral drugs: a global warning. Top Antivir Med. 2014 Jan;21(5):165-8. PMID 24531557
- [Result] Avihingsanon A, Jitmitraparp S, Tangkijvanich P, Ramautarsing RA, Apornpong T, Jirajariyavej S, Putcharoen O, Treeprasertsuk S, Akkarathamrongsin S, Poovorawan Y, Matthews GV, Lange JM, Ruxrungtham K; HIV-NAT125 study team. Advanced liver fibrosis by transient elastography, fibrosis 4, and alanine aminotransferase/platelet ratio index among Asian hepatitis C with and without human immunodeficiency virus infection: role of vitamin D levels. J Gastroenterol Hepatol. 2014 Sep;29(9):1706-14. doi: 10.1111/jgh.12613. PMID 24730732
- [Result] Wattanakul T, Avihingsanon A, Manosuthi W, Punyawudho B. Population pharmacokinetics of nevirapine in Thai HIV-infected patients. Antivir Ther. 2014;19(7):651-60. doi: 10.3851/IMP2741. Epub 2014 Feb 6. PMID 24504545
- [Result] Durier N, Ananworanich J, Apornpong T, Ubolyam S, Kerr SJ, Mahanontharit A, Ferradini L, Ruxrungtham K, Avihingsanon A. Cytomegalovirus viremia in Thai HIV-infected patients on antiretroviral therapy: prevalence and associated mortality. Clin Infect Dis. 2013 Jul;57(1):147-55. doi: 10.1093/cid/cit173. Epub 2013 Mar 19. PMID 23511301
- [Result] Praditpornsilpa K, Avihingsanon A, Chaiwatanarat T, Chaiyahong P, Wongsabut J, Ubolyam S, Chulakadabba A, Avihingsanon Y, Ruxrungtham K, Tunsanga K, Eiam-Ong S, Phanuphak P. Comparisons between validated estimated glomerular filtration rate equations and isotopic glomerular filtration rate in HIV patients. AIDS. 2012 Sep 10;26(14):1781-8. doi: 10.1097/QAD.0b013e328356480d. PMID 22713478
- [Result] Kerr SJ, Duncombe C, Avihingsanon A, Ananworanich J, Boyd M, Sopa B, Medtech B, Chuenyam T, Cooper DA, Lange JM, Phanuphak P, Ruxrungtham K. Dyslipidemia in an Asian population after treatment for two years with protease inhibitor-containing regimens. J Int Assoc Physicians AIDS Care (Chic). 2007 Mar;6(1):36-46. doi: 10.1177/1545109706295946. PMID 17329503
- [Result] Avihingsanon A, Avihingsanon Y, Darnpornprasert P, Kerr S, Ungsedhapand C, Duncombe C, Ubolyam S, Ruxrungtham K, Phanuphak P. High prevalence of indinavir-associated renal complications in Thai HIV-infected patients. J Med Assoc Thai. 2006 Aug;89 Suppl 2:S21-7. PMID 17044450
- [Derived] Gatechompol S, Lutter R, Vaz FM, Ubolyam S, Avihingsanon A, Kerr SJ, van Leth F, Cobelens F. The plasma kynurenine-to-tryptophan ratio as a biomarker of tuberculosis disease in people living with HIV on antiretroviral therapy: an exploratory nested case-control study. BMC Infect Dis. 2024 Apr 2;24(1):372. doi: 10.1186/s12879-024-09258-4. PMID 38565993
- [Derived] Wattanachanya L, Sunthornyothin S, Apornpong T, Lwin HMS, Kerr S, Gatechompol S, Han WM, Wichiansan T, Siwamongsatham S, Chattranukulchai P, Chaiwatanarat T, Avihingsanon A; HIV-NAT 207/006 study team. Bone mineral density among virologically suppressed Asians older than 50 years old living with and without HIV: A cross-sectional study. PLoS One. 2022 Nov 21;17(11):e0277231. doi: 10.1371/journal.pone.0277231. eCollection 2022. PMID 36409740
- [Derived] Gatechompol S, Avihingsanon A, Apornpong T, Han WM, Kerr SJ, Ruxrungtham K. Efficacy and improvement of lipid profile after switching to rilpivirine in resource limited setting: real life clinical practice. AIDS Res Ther. 2019 Apr 5;16(1):7. doi: 10.1186/s12981-019-0222-6. PMID 30953533
- [Derived] Han WM, Apornpong T, Kerr SJ, Hiransuthikul A, Gatechompol S, Do T, Ruxrungtham K, Avihingsanon A. CD4/CD8 ratio normalization rates and low ratio as prognostic marker for non-AIDS defining events among long-term virologically suppressed people living with HIV. AIDS Res Ther. 2018 Sep 27;15(1):13. doi: 10.1186/s12981-018-0200-4. PMID 30261902
- [Derived] Punyawudho B, Thammajaruk N, Thongpeang P, Matthews G, Lewin SR, Burger D, Ruxrungtham K, Avihingsanon A. Population pharmacokinetics of tenofovir in HIV/HBV co-infected patients. Int J Clin Pharmacol Ther. 2015 Nov;53(11):947-54. doi: 10.5414/CP202386. PMID 26308175
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org